CLINICAL TRIAL: NCT06408532
Title: The Evaluation of the Efficacy and Safety of Switching to Once-daily IDegLira in Patients With Type 2 Diabetes Receiving Premixed Insulin Therapy, a Multi-center, Randomized Control Trial
Brief Title: The Efficacy and Safety of Insulin Degludec/Liraglutide Combination (IDegLira) in Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Liu, Associate Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD 2023-02
Record Dates: First submitted 2024-04-25; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Premixed insulin dose optimization group (Active Comparator): The participants in this group will get optimized insulin dosage adjustment on premixed insulin.
  Interventions: Drug: Premixed insulin
- IDegLira once daily injection group (Experimental): The participants in this group will switch from premixed insulin to IDegLira once daily injection therapy.
  Interventions: Drug: IDegLira

INTERVENTIONS:
Drug: IDegLira — The participants in this group will be switched to IDegLira once daily injection therapy.
  Arms: IDegLira once daily injection group
Drug: Premixed insulin — The participants in this group will be have optimized premixed insulin regimen.
  Arms: Premixed insulin dose optimization group

SUMMARY:
The study aims to evaluate the efficacy and safety of IDegLira in type 2 diabetes who have failed premixed insulin therapy. The study plans to enroll 256 participants with inadequate glycemic control despite twice-daily subcutaneous injections of premixed insulin and metformin. Participants will be randomly assigned to either the premixed insulin dose optimization group (control group) or IDegLira once daily group, and the difference in change in glycated hemoglobin levels from baseline to 16 weeks of treatment will be assessed between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for ≥3 months. Meets the diabetes diagnostic criteria established by the World Health Organization (WHO) in 1999.
* Age ≥18 years, regardless of gender.
* Body mass index ≥23.0 kg/m^2.
* HbA1c ≥7.5% and ≤11.0% at screening.
* Concurrently taking metformin, with a metformin dose ≥1500 mg/day or the maximum tolerated dose (not less than 1000 mg/day), and may be combined with oral sodium-glucose cotransporter-2 inhibitors, thiazolidinediones, or alpha-glucosidase inhibitors. Combination oral medications must be at a stable dose for ≥8 weeks and continued during the study period.
* For 8 weeks prior to screening, has been on a stable, regular regimen of premixed human insulin (including premixed insulin analogs) administered subcutaneously twice daily, with a total daily insulin dose of 15-50 units, in addition to diet and exercise control.
* Has signed the informed consent form.
* Willing and able to self-monitor blood glucose (SMBG) and record the diary card on time.
* Fully understands the study purpose and can communicate well with the investigator, and can understand and comply with all requirements of this study.

Exclusion Criteria:

* Subjects who have previously tested positive for diabetes autoantibodies (including anti-glutamic acid decarboxylase antibodies, anti-islet cell antibodies, anti-insulin antibodies, anti-zinc transporter 8 antibodies, and anti-protein tyrosine phosphatase antibodies).
* Fasting C-peptide level ≤0.6 ng/mL.
* Used a glucagon-like peptide-1 (GLP-1) receptor agonist within the 3 months prior to screening.
* Concomitant use of sulfonylureas, glinides, and dipeptidyl peptidase-4 inhibitors within the 3 months prior to screening.
* History of medullary thyroid carcinoma, multiple endocrine neoplasia type 2, or a family history of these conditions.
* History of acute/chronic pancreatitis.
* Experienced a serious gastrointestinal disease (such as active ulcer) or underwent gastrointestinal surgery (except appendectomy or cholecystectomy) or had clinically significant gastric emptying abnormalities (such as pyloric obstruction, gastroparesis) or long-term use of medications that directly affect gastrointestinal motility, or deemed unsuitable for the study by the investigator within the 3 months prior to screening.
* Concurrent severe diseases, including but not limited to severe cardiovascular, cerebrovascular, hepatic, or renal diseases, or severe diabetes-related complications, and deemed unsuitable for the study by the investigator.
* Pregnant or breastfeeding female subjects, or subjects (including male subjects' female partners) with plans for pregnancy or sperm/egg donation within 3 months after the last dose, or unwilling to use at least one effective contraceptive method or device.
* Unwilling to wear an invasive monitoring device.
* Clear reasons that prevent the use of continuous glucose monitoring (CGM), such as severe allergy or skin conditions, and deemed unsuitable for the study by the investigator.
* Subjects with skin lesions, scarring, redness, infection, or edema at the sensor application site that may affect the accuracy of sensor placement or interstitial glucose measurement.
* Received long-term (continuous or cumulative ≥7 days) treatment with systemic corticosteroids or growth hormone that may affect blood glucose within 1 month prior to screening.
* History of malignancy within the past 3 years, excluding basal cell carcinoma, squamous cell carcinoma, and any in situ cancers.
* Participated in another drug or medical device clinical trial (except for registry studies) within the 3 months prior to screening.
* Presence of severe psychiatric disorders or language barriers, unwilling or unable to fully understand and cooperate.
* Experienced diabetic ketoacidosis (DKA), hyperosmolar hyperglycemic state (HHS), or lactic acidosis (LAD) within the 3 months prior to screening.
* Fasting triglycerides >5.65 mmol/L (can be retested within one week) at screening.
* History of alcohol or drug abuse (more than 14 units of alcohol per week [1 unit = 360 mL of 5% beer, or 45 mL of 40% spirits, or 150 mL of 12% wine]).
* Known or suspected allergy to GLP-1 class drugs or excipients.
* Any other reason deemed by the investigator to make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | From baseline to the end of the study (week 0-week 14 ± 7days).
  The change in glycated hemoglobin levels from baseline at the end of the study

SECONDARY OUTCOMES:
Time in Range (TIR, 3.9-10.0 mmol/L) obtained from Continuous Glucose Monitoring (CGM) | CGM data collected at the end of the study (week 14 ± 7days).
Time in Tight Range (TTIR, 3.9-7.8 mmol/L) | CGM data collected at the end of the study (week 14 ± 7days).
Glucose Management Indicator (GMI) | CGM data collected at the end of the study (week 14 ± 7days).
Prolonged Hypoglycemic Events (defined as glucose <3.9 mmol/L for ≥120 minutes, with event ending when glucose ≥3.9 mmol/L for ≥15 minutes) | CGM data collected at the end of the study (week 14 ± 7days).
Prolonged Hyperglycemic Events (defined as glucose >13.9 mmol/L for ≥120 minutes, with event ending when glucose ≤10 mmol/L for ≥15 minutes) | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with TIR (3.9-10 mmol/L) >70% | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with ≥5% improvement in TIR (3.9-10 mmol/L) from baseline at study end. | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with ≥10% improvement in TIR (3.9-10 mmol/L) from baseline at study end | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with Time Below Range (TBR, <3.9 mmol/L) <4% | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with Time Below Range (TBR, <3.0 mmol/L) <1% | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with Time Above Range (TAR, >10.0 mmol/L) <25% | CGM data collected at the end of the study (week 14 ± 7days).
Percentage of patients with Time Above Range (TAR, >13.9 mmol/L) <5% | CGM data collected at the end of the study (week 14 ± 7days).
The frequency of confirmed hypoglycemia | From baseline to the end of the study (week 0-week 14 ± 7days).
  Having symptoms of hypoglycemia and a fingerstick blood glucose measurement of <4mmol/L.
Frequency of confirmed nocturnal hypoglycemia | From baseline to the end of the study (week 0-week 14 ± 7days).
  Confirmed hypoglycemia occurring at night
Frequency of severe hypoglycemia | From baseline to the end of the study (week 0-week 14 ± 7days).
  hypoglycemia that the individual cannot self-treat and requires assistance from another person
Change in body weight from baseline | From baseline to the end of the study (week 0-week 14 ± 7days).
Change in waist circumference from baseline | From baseline to the end of the study (week 0-week 14 ± 7days).
Short-Form Health Survey (SF-36) | At the end of the study (week 14 ± 7days).
  A score ranging from 0 to 100. Higher scores indicate better health status.
Diabetes Treatment Satisfaction Questionnaire (DTSQs) ④ Exploratory Evaluation Indicators | At the end of the study (week 14 ± 7days).
  The DTSQs is composed of six items and scored on seven-point response scales ranging from "very satisfied" (assigned a score of 6) to "very unsatisfied" (assigned a score of 0). Higher DTSQs scores indicate greater satisfaction with treatment (range 0 to 36).
Changes in the Ambulatory Glucose Profile (AGP) graph obtained from CGM | From baseline to the end of the study (week 0-week 14 ± 7days).

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) could be accessed with proper reason from the PI.